CLINICAL TRIAL: NCT03333265
Title: The Effect of Berberine Hydrochloride in Familial Adenomatous Polyposis:a Prospective, Randomized, Double Blind, Placebo-controlled, Multicenter Clinical Trial
Brief Title: Primary Chemoprevention of Familial Adenomatous Polyposis With Berberine Hydrochloride
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, xiaohua li, Director of colorectal surgery center, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: XJLL 2016 017
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Colorectal Adenomas

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 100mg Berberine hydrochloride group (Experimental): Berberine hydrochloride 100mg tablet by mouth, two times per day for 6 months
  Interventions: Drug: 100mg Berberine hydrochloride
- 300mg Berberine hydrochloride group (Experimental): Berberine hydrochloride 300mg tablet by mouth, two times per day for 6 months
  Interventions: Drug: 300mg Berberine hydrochloride
- Placebo oral tablets (Placebo Comparator): identical-appearing placebo tablets by mouth, two times per day for 6 months
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: 100mg Berberine hydrochloride — patients take the Berberine hydrochloride 100mg tablet by mouth, 2 times a day with 6 months
  Other Names: 100mg Berberine hydrochloride tablet ("Sine Tianping")
  Arms: 100mg Berberine hydrochloride group
Drug: 300mg Berberine hydrochloride — patients take the Berberine hydrochloride 300mg tablet by mouth, 2 times a day with 6 months
  Other Names: 300mg Berberine hydrochloride tablet ("Sine Tianping")
  Arms: 300mg Berberine hydrochloride group
Drug: Placebo Oral Tablet — patients take mmic Berberine hydrochloride tablet by mouth, 2 times a day with 6 months
  Other Names: Placebo (for Berberine hydrochloride)
  Arms: Placebo oral tablets

SUMMARY:
In recent years, Berberine hydrochloride has been reported to inhibit cancer cell proliferation and to be cytotoxic towards cancer cells. Patients with familial adenomatous polyposis have a nearly 100 percent risk of colorectal cancer. The aim of this study is to investigate the chemopreventive effects Berberine hydrochlorid on the regression of colorectal adenomas.

DETAILED DESCRIPTION:
Familial adenomatous polyposis is an autosomal dominant syndrome caused by a germ-line mutation of the adenomatous polyposis coli (APC) gene located at chromosome 5q21. The disorder is characterized by the development of hundreds of colorectal adenomas during adolescence. Colorectal cancer will develop in nearly all affected persons by the sixth decade of life if prophylactic colectomy is not performed. Because the adenoma-to-carcinoma sequence in familial adenomatous polyposis resembles sporadic colon carcinogenesis, studies of familial adenomatous polyposis may contribute to the prevention of sporadic adenomas and colon cancer.

BBR, an isoquinoline alkaloid, is a natural compound in numerous Chinese herb plants such as Berberisaristata, Coptischinensis, Coptis rhizome, etc. In recent years, Berberine hydrochloride has been reported to inhibit cancer cell proliferation and to be cytotoxic towards cancer cells. The aim of this study is to investigate the regression effect of Berberine hydrochloride on the colorectal adenomas in patients with familial adenomatous polyposis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years
* Patients with familial adenomatous polyposis, who had not had their entire colorectum removed, and who had five or more polyps 2 mm or more in diameter that could be assessed endoscopically
* All potential subjects received genetic counseling before undergoing genetic testing for APC gene mutations.
* Eligible subjects had a disease-causing mutation of the APC gene but had no endoscopically detectable colorectal adenomatous polyps and no history of colonic surgery

Exclusion Criteria:

* Patients who are hypersensitive or intolerant to the drugs
* Patients who had a history of colectomy or colectomy anticipated within 8 months after randomization
* Patients with abnormal results of serum laboratory tests (a white-cell count of less than 4000 per cubic millimeter, a platelet count of less than 100,000 per cubic millimeter, a blood urea nitrogen level of more than 25 mg per deciliter (8.9 mmol per liter), a serum creatinine level of more than 1.5 mg per deciliter (132.6 µmol per liter))
* Patients with diabetes mellitus, severe renal disease or cardiovascular disease (defined by a New York Heart Association functional classof III or IV)
* Patients with hypercalcemia or urolithiasis
* Patients with hemolytic anemia and glucose -6- phosphate dehydrogenase deficiency
* Patients had clinically obvious narcotic or alcohol dependence during the previous 6 months
* Patients had used NSAIDs including aspirin at any dose on 3 or more days per month during each of the 3 months before enrollment or for a period of 36 days in the previous year; or had a history of stroke, transient ischemic attacks, angina, myocardial infarction, or atherosclerotic peripheral vascular disease
* Pregnant women, women during breast-feeding period, or women with expect pregnancy
* Patients with a history of subtotal gastrectomy or partial bowel resection
* Patients who are not able to cooperate
* Individual who are involved in designing, planning or performing this clinical trial
* Patients with medical conditions who are not appropriate to participate the study
* Patients with any condition that could be worsened by supplemental Berberine hydrochloride

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Cumulative the numbers and diameters of those colorectal adenomas during Berberine hydrochloride or placebo treatment in patients with familial adenomatous polyposis | From baseline to 6 months.
  The primary objective of this study is to investigate the number and diameters of colorectal polyps after Berberine hydrochloride or placebo intervention. To ascertain that the same area was scored at base line and at month 6, polyps were counted in pairs of photographs. One investigator, other than the endoscopist, who did not know the treatment, performed the scoring. Videotapes were used to resolve ambiguities and confirm polyp counts. The diameter of those colorectal adenomas was measured in millimeters with a graduated scale passed through the colonoscopy biopsy channel.

CONTACTS AND LOCATIONS:
Overall Officials: Weizhong Wang, MD,PH.D, Principal Investigator — Xijing digestive surgery center
Locations (1):
- Li, Xi'an, Shaanxi, China